CLINICAL TRIAL: NCT05779176
Title: Safety and Efficacy of Therapeutic Hypothermia in Acute Ischemic Stroke Patients Treated With Mechanical Thrombectomy: a Prospective, Randomized, Controlled Clinical Study
Brief Title: Safety and Efficacy of Therapeutic Hypothermia in Acute Ischemic Stroke
Acronym: THIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, LiqunYang, archiater, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA-2022-180
Record Dates: First submitted 2023-02-23; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Ischemic
Keywords: Therapeutic hypothermia, AIS, Neurological function prognosis
MeSH Terms: conditions — Ischemic Stroke | interventions — Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: Safety and efficacy of therapeutic hypothermia in acute ischemic stroke (AIS) patients treated with Intravascular thrombectomy is a prospective, multi-center, randomized, parallel-group interventional study.
Masking Description: This trial is open labeled, the treatment allocation is known to the treating physicians and the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normothermia arm (No Intervention): Patients randomized to normothermia will be maintained at 36-37°C during the entire study period.
- Therapeutic hypothermia arm (Experimental): Patients assigned to TH will receive intravascular temperature management to achieve the target temperature of 34-35 °C
  Interventions: Procedure: Therapeutic hypothermia

INTERVENTIONS:
Procedure: Therapeutic hypothermia — The study intervention is therapeutic hypothermia. After intubation, patients assigned to therapeutic hypothermia will receive central venous catheterization through right jugular vein or femoral vein depending on the cooling application and the unique needs, a flexible catheter will be inserted and iced saline was circulated through the multiple balloons of the catheter in a closed-loop design to induce therapeutic hypothermia. This system also has a hydrophilic coating with heparin and a triple-lumen central venous catheter to satisfy the need of fluid or drug infusion, blood draw and central venous pressure monitoring. After central venous catheterization, patients assigned to TH will receive intravascular temperature management to achieve the target temperature of 34-35 °C.
  Arms: Therapeutic hypothermia arm

SUMMARY:
Therapeutic hypothermia (TH) in stroke has demonstrated robust neuroprotection in animals especially after ischemia-reperfusion injury, but its safety and efficacy remain controversial. The investigators propose this trial to study the clinical and radiological effects of therapeutic hypothermia in acute ischemic stroke patients treated with intravascular thrombectomy (IVT).

DETAILED DESCRIPTION:
The study intervention is therapeutic hypothermia. After intubation, patients assigned to therapeutic hypothermia will receive central venous catheterization through right jugular vein or femoral vein depending on the cooling application and the unique needs, a flexible catheter will be inserted and iced saline will be circulated through the multiple balloons of the catheter in a closed-loop design to induce therapeutic hypothermia. This system also has a hydrophilic coating with heparin and a triple-lumen central venous catheter to satisfy the need of fluid or drug infusion, blood draw and central venous pressure monitoring. After central venous catheterization, patients assigned to TH will receive intravascular temperature management to achieve the target temperature of 34-35 °C, which is superior to surface methods in cooling performance in terms of faster rate of cooling, shorter induced cooling time, precise control during maintenance. Thereafter, hypothermia will be maintained for 24 hrs from the start of hypothermia. The patients will be rewarmed slowly at a rate of no greater than 0.5 °C every 4 h. What's more, patients in TH group will execute anti-shivering protocol during awaking and extubation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-85 years(inclusive);
2. Patients have clinical signs consistent with acute ischemic stroke,
3. Patients with acute large vessel occlusion including internal carotid artery and middle cerebral artery M1 and M2 demonstrated by CTA，MRA or DSA
4. The possibility to receive arterial thrombus removal treatment （within6 or24 hr of large vessel occlusion ）;
5. Provide the informed consent form of the patient or the patient's agent.

Exclusion Criteria:

1. Coma or altered vigilance defined as a score ≥2 on the level of consciousness 1A subscale of the NIHSS.
2. Associated cerebral hemorrhage.
3. There is dysfunction before the onset, mRS score >= 2 points;
4. Accompanied by severe comorbidities (such as severe cardiopulmonary insufficiency, the expected survival period of advanced malignant tumors is less than 90 days);
5. Multi-mode CT/MRI examination of the corresponding contrast agent use contraindications (such as contrast agent allergy, etc.);
6. Women during pregnancy or lactation;
7. Patients currently participating in other clinical research trials;
8. Other conditions judged by the investigator as not suitable for inclusion in the clinical study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Neurological function prognosis | 90±14 days post-operation
  the score on the modified Rankin Scale, seven grades ranked from 0 to 6, higher scores mean worse outcome

SECONDARY OUTCOMES:
Ratio of mRS score 2 or less | 90±14 days post-operation
  the ratio of modified Rankin Scale score 2 or less, modified Rankin Scale has seven grades ranked from 0 to 6, higher scores mean worse outcome
Incidence of intracranial hemorrhage and symptomatic intracranial hemorrhage | 24-72 hours post-operation
  Radiological examination（CT or MRI）
Target vascular recanalization rate | 24-72 hours post-operation
  Cerebral angiography
NIHSS score | 7 days post-operation
  The score of National Institute of Health stroke scale, NIHSS score ranked from 0 to 42, higher scores mean a worse neurological outcome
Final infarct volume | 7 days post-operation
  CT scan
Death in hospital & within 90 days | Within 90 days after admission
  Death in 90 days
The incidence of adverse event | Within 7 days post-operation
  Surgery-related complications: vascular perforation, arterial dissection, and distal embolization；Incidence of pneumonia within 7 days; Incidence of deep vein thrombosis within 7 days
Adverse events of hypothermia and rewarming | Within 24 hours post-operation
  arrhythmia (atrial fibrillation, ventricular fibrillation), hypokalemia, Chilblains or pressure ulcers; Rewarming shock and hyperkalemia

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Yang, Ph.D., Principal Investigator — Renji Hospital, Shanghai Jiao Tong University School of Moedicine
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China

REFERENCES:
- [Background] Mendelson SJ, Prabhakaran S. Diagnosis and Management of Transient Ischemic Attack and Acute Ischemic Stroke: A Review. JAMA. 2021 Mar 16;325(11):1088-1098. doi: 10.1001/jama.2020.26867. PMID 33724327
- [Background] Feigin VL, Norrving B, Mensah GA. Global Burden of Stroke. Circ Res. 2017 Feb 3;120(3):439-448. doi: 10.1161/CIRCRESAHA.116.308413. PMID 28154096
- [Background] Chio CC, Kuo JR, Hsiao SH, Chang CP, Lin MT. Effect of brain cooling on brain ischemia and damage markers after fluid percussion brain injury in rats. Shock. 2007 Sep;28(3):284-90. doi: 10.1097/SHK.0b013e3180311e60. PMID 17529907
- [Background] Hynson JM, Sessler DI, Moayeri A, McGuire J. Absence of nonshivering thermogenesis in anesthetized adult humans. Anesthesiology. 1993 Oct;79(4):695-703. doi: 10.1097/00000542-199310000-00010. PMID 8214747
- [Background] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793